CLINICAL TRIAL: NCT02625493
Title: Patient Preferences for Radial Versus Femoral Vascular Access Options by Coronary Angiography and Intervention
Brief Title: Patient Preference for Radial Versus Femoral Vascular Access
Acronym: PREVAS
Status: Completed | Type: Observational
Sponsor: Thorax Centrum Twente (Other)
Collaborators: Foundation of Cardiovascular Research and Education Enschede (Other)
Responsible Party: Principal Investigator, Clemens von Birgelen, MD, PhD, Thorax Centrum Twente
Other Study IDs: Prevas-v2
Record Dates: First submitted 2015-11-30; First posted 2015-12-09 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Coronary Artery Disease
Keywords: Percutaneous coronary intervention; Patient Preference; Radial access; Femoral access; Coronary angiography; Shared decision making
MeSH Terms: conditions — Coronary Artery Disease; Patient Preference | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- study population: All patients who underwent elective coronary procedures belonged to the one group, they received standard care without any additional interventions, but were asked to fill in a questionnaire.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaire containing a Best-worst Scaling scenario

SUMMARY:
The purpose of this study is to determine the preference of patients regarding the vascular access site in future coronary procedures. We hypothesize that patients prefer the lesser invasive procedure via radial access.

DETAILED DESCRIPTION:
Rationale: To explore patient preference for vascular access site in percutaneous coronary procedures, by assessing the perceived importance of benefits and risks of both transradial access and transfemoral access. In addition, direct preference for vascular access and preference for shared decision-making were evaluated.

Objective: To investigate the patient preference of vascular access -transradial versus transfemoral- in future percutaneous coronary procedures, by use of the Best-Worst Scaling.

Study design: Single-center, prospective, observational registry

Study population: A consecutive series of patients, who between June and August 2014, underwent elective coronary procedures at Thoraxcentrum Twente in Enschede.

Intervention: All subjects will receive a questionnaire containing basic baseline questions and a best-worst scaling scenario in which they were asked to indicate the most and least desirable characteristics of the vascular access approach.

Furthermore, their direct preference was asked and to which extent they preferred to participate in the decision-making process regarding the choice for vascular access route in future percutaneous coronary procedures.

Main study endpoints:

* The primary endpoint is the patient preference on specific treatment characteristics with regard to vascular access in coronary procedures.
* Secondary endpoints include

  1. direct patient preference for transradial access or transfemoral access
  2. the valuation of participation in decision-making on the choice of vascular access together with the interventional cardiologist.

ELIGIBILITY:
Inclusion Criteria:

* All patients who undergoing an elective coronary procedure at Thoraxcenteum Twente in the period of June 2014 until August 2014

Exclusion Criteria:

* Language barrier

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A consecutive series of patients, who between June and August 2014, underwent elective coronary procedures at Thoraxcentrum Twente in Enschede.
Sampling Method: Non-Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2014-06; Primary Completion 2014-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
The best and worst treatment characteristics of transradial and transfemoral access, by using a software-generated Best-Worst Scaling Questionnaire - case 2 | 30 days
  Best-Worst Scaling Questionnaire will be used to assess which treatment characteristics patients find most and least desirable in percutaneous coronary procedures performed via transradial and transfemoral access.

OTHER OUTCOMES:
Number of times that patients prefer transradial in future percutaneous coronary procedure, when given a discrete choice via a questionnaire. | 30 days
  When given the discrete choice, which access site patients would prefer in future percutaneous coronary procedures.
Percentage of patients that wants to be directly involved in the decision-making process when making the choice for access site in future coronary procedures, by use of a questionnaire. | 30 days
  The valuation of participation in decision-making on the choice of vascular access together with the interventional cardiologist

CONTACTS AND LOCATIONS:
Overall Officials: Harald Verheij, Study Director — research manager
Locations (1):
- Medisch Spectrum Twente, Enschede, Netherlands

REFERENCES:
- [Derived] Kok MM, Weernink MGM, von Birgelen C, Fens A, van der Heijden LC, van Til JA. Patient preference for radial versus femoral vascular access for elective coronary procedures: The PREVAS study. Catheter Cardiovasc Interv. 2018 Jan 1;91(1):17-24. doi: 10.1002/ccd.27039. Epub 2017 May 4. PMID 28470994